CLINICAL TRIAL: NCT06892197
Title: Comparing Hydrocortisone and Prednisolone for Community Acquired Pneumonia (CAP)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen Respiratory Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MineraloCAP
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Community Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methylprednisolone; Pharmaceutical Preparations; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomized controlled trial. It consists of two arms, in which patients will be randomized to receive treatment with either Hydrocortisone or Prednisolone.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Hydrocortisone. (Active Comparator): This arm will recieve a dose of 200 mg of Hydrocortisone intravenously once daily for five days.
  Interventions: Drug: hydrocortisone
- Treatment with Methylprednisolone (Active Comparator): This arm will recieve a dose of 40 mg of Methylprednisolone intravenously once daily for five days.
  Interventions: Drug: Methylprednisolone (drug)

INTERVENTIONS:
Drug: Methylprednisolone (drug) — ATC code: H02AB06. Can be changed to Prednisolone 50 mg orally.
  Arms: Treatment with Methylprednisolone
Drug: hydrocortisone — ATC-code: H02AB09. Can be changed to 50 mg x 4 daily orally if appropriate.
  Arms: Treatment with Hydrocortisone.

SUMMARY:
The goal of this cluster randomized controlled trial is to determine the optimal treatment for community aquired pneumonia (CAP). The study compares the effects and side effects of hydrocortisone and prednisolone in patients above 18 years old diagnosed with severe CAP. The main question is whether there is a difference in all cause mortality within thirty days.

Participants will be randomized to receive treatment with either hydrocortisone or prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of severe CAP for who the physician in charge decides for corticosteroid therapy for severe CAP.

Exclusion Criteria:

* Admitted >24 h
* Pregnant or breastfeeding women
* Active tuberculosis or fungal infection
* Pneumonia caused by influenza
* Intolerance to either study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 90 days
All-cause infections | 90 days
Need for vasopressor treatment | 30 days
Need for mechanical ventilation | 30 days
Admission to ICU | 30 days
Daily amount of insulin administered to the patient by day 7 or discharge from hospital | 7 days
Gastrointestinal bleeding | 30 days
Blood glucose levels | 7 days
  Measured at day 3 and day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Stæhr Jensen, MD, PHD, Study Director — COP:RESP

IPD SHARING:
Plan to Share IPD: Undecided
This has not yet been decided.